CLINICAL TRIAL: NCT06115330
Title: The Effectiveness of Battlefield Acupuncture (BFA) With Standard Therapy Compared With Standard Therapy in Gynecological Cancer Pain
Brief Title: The Effectiveness of Battlefield Acupuncture (BFA) With Standard Therapy in Gynecological Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Alvita Ratnasari, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-06-0971
Record Dates: First submitted 2023-08-29; First posted 2023-11-03 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Gynecologycal Cancer; Cancer Related Pain; Cancer Pain
Keywords: Battlefield acupuncture; Ear acupuncture; Cancer pain; Gynecologycal cancer pain; Quality of life
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ear Acupuncture with Standard Medical Therapy (Experimental): The intervention group was give a press needle acupuncture with standard medical therapy for gynecological cancer pain
  Interventions: Device: Press Needle Acupuncture
- Standard Medical Therapy (No Intervention): The control group was given standard medical therapy for gynecological cancer pain

INTERVENTIONS:
Device: Press Needle Acupuncture — Ear acupuncture using Pyonex press needles were installed with a diameter of 0.17mm, 0.9mm deep. The needles were retained for three days and stimulated at the installation site of the patch needle by means of pressure on the acupuncture point ears that have been attached needles on both sides, 1 minute at each point, four times a day, for 3 consecutive days and the patch was removed on the 3rd day
  Arms: Ear Acupuncture with Standard Medical Therapy

SUMMARY:
Pain is one of the most important symptoms of cancer patients, with nearly 40% of all cancer patients experiencing moderate to severe pain. Gynecological oncology patients on palliative care have a chief complaint of pain or significant nausea/vomiting, contrary to the patient's initial complaints on admission such as fever, infection, dyspnea, changes, altered consciousness, bleeding, pancytopenia. Strong recommendations by WHO regarding the use of non-steroidal anti-inflammatory drugs (NSAIDs), paracetamol and opioids either alone or in combination in adults, including the elderly and adolescents with cancer-related pain in the early stages, pain relief depending on clinical judgment and severity to achieve pain treatment which is fast and safe. Ear acupuncture is a simple and safe method that can be used alone or in combination with other forms of medical care, which is effective in treating a variety of conditions as well as painful conditions. Based on the previous 2020 systematic review regarding ear acupuncture in its benefits in cancer pain, it was stated that ear acupuncture was effective in treating pain in cancer patients with moderate pain levels, effective for reducing pain scores, faster onset, and longer duration of analgesics. Ear acupuncture is also more effective when compared to standard therapy without acupuncture, so it can be used as an additional modality for cancer pain. Currently there is no research on the effectiveness of BFA ear acupuncture therapy in the treatment of gynecological cancer pain to treat it based on the consistency of point selection, so it is necessary to conduct research on the effectiveness of BFA ear acupuncture therapy in the treatment of gynecological cancer pain.

This study aim to analyze the effectiveness of BFA ear acupuncture therapy plus standard therapy on pain intensity (VAS score), changes in analgesic dose, and quality of life (EORTC QLQ C-30 score) in patients with gynecological cancer pain compared to standard therapy alone.

DETAILED DESCRIPTION:
This study was conducted using a single blinded randomized control clinical trial design in 58 female patients who are hospitalized aged 18-65 years, have a diagnosis of gynecological cancer, with a VAS score≥4 caused by tumor, before or during a therapeutic process (radiation therapy, chemotherapy, or after surgery), agree to participate in the study, sign the informed consent form who were randomized into 2 groups, namely group I BFA ear acupuncture with standard therapy and group 2 standard therapy, the acupuncture points used were placed at points MA-IT1 Cingulate Gyrus, MA-AT2 Thalamus, MA-H2 Omega 2, MA-H1 Point Zero, MA-TF1 Shenmen on both sides of the ear using Pyonex needles were placed with a diameter of 0.17mm, depth of 0.9mm. the pyonex press needle. were retained for three days The outcome assessed were pain intensity using the VAS, changes in analgesic dose, and quality of life with the EORTC QLQ C-30 questionnaire, which was assessed on the day before starting therapy, the first day, the second day, the third day, the fifth day and the seventh day

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with gynecological cancer.
* Women over 18 years to 65 years
* Subjects experiencing pain in cancer, with VAS ≥4, namely pain that caused by

  * tumors,
  * before or during a therapeutic process (radiation therapy, chemotherapy or postoperatively).
  * side effect or the result of toxicity of cancer treatment.
* Willing to participate in this research and sign informed consent

Exclusion Criteria:

* The patient has a medical emergency / hemodynamically unstable.
* Uncooperative patients, with serious psychological disorders, no currently undergoing psychiatric treatment, aggressive behavior, no allow for acupuncture.
* Patients with blood clotting disorders, with platelets <50.000114 and in neutropenic condition with <1000 neutrophils. 114
* The patient has an allergy to stainless steel acupuncture needles.
* Wounds at the acupuncture point puncture sites, skin infections in the ears. On patients with eczema on the ears, external otitis or psoriasis.
* There is a tumor in the area that will be stabbed and stimulated in the stomach pregnant women, close to the heart, or in the area of the carotid sinus lymphedema, insertion into the prosthesis.
* Patients with heart rhythm disorders.
* The patient uses a pace maker.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Pain Severity with Visual Analog Scale | Before treatment, After treatment in day 1, day 2, day 3, day 5 and day 7
  Rating scale for measuring pain, where the minimum value is 0 = no pain, and the maximum value is 100 = severe pain. A higher scale means worse outcomes.
  assessment used to assess intensity of certain sensations and feelings, like pain.

SECONDARY OUTCOMES:
Quality of Life with European Organisation for Research and Treatment of Cancer Quality of Life C30 | before treatment and 7 day after treatment
  European Organisation for Research and Treatment of Cancer Quality of Life C30, that include two item of review functional scale and the global health scale both scale the higher the score the outcome will be better
Analgetic Usage | Before treatment, After treatment in day 1, day 2, day 3, day 5 and day 7
  Analgetic used during the treatment measured in miligram

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia
Locations (3):
- Indonesia (3):
  - Fatmawati Hospital, Jakarta, DKI Jakarta
  - Persahabatan Hospital, Jakarta, DKI Jakarta
  - Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: No